CLINICAL TRIAL: NCT03919708
Title: Deploying Retinal Birefringence Imaging in to the Clinic for Pediatric Vision Screening
Brief Title: Amblyopia and Strabismus Detection Using Retinal Birefringence Imaging
Acronym: RBI
Status: Withdrawn | Type: Observational
Why Stopped: Funding expired
Sponsor: Rebiscan, Inc. (Industry)
Collaborators: Retina Foundation of the Southwest (Other)
Responsible Party: Sponsor
Other Study IDs: rebiscan_RBI_RFSW
Record Dates: First submitted 2019-04-16; First posted 2019-04-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Amblyopia; Strabismus
MeSH Terms: conditions — Amblyopia; Strabismus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Enriched Population: Children between the ages of 2-8 who present to an eye clinic. Eligible and recruited children will be scanned with a PVS device and an RBI device, and then be provided with a full, gold standard eye exam by a pediatric ophthalmologist. All scans and exam should be performed within a single visit. Scans should take no longer than 20 seconds each, and ophthalmic exam should take approximately 30 minutes.
  Interventions: Device: Retinal Birefringence Imager
- Unenriched Population: Children between the ages of 2-8 who present to a general pediatric clinic, with no history of eye disorders or amblyopia. Eligible and recruited children will be scanned with a PVS device and an RBI device, and then be provided with a full, gold standard eye exam by a pediatric ophthalmologist. All scans will be performed at a single visit, but the exam may require a follow up visit, depending on the availability of a pediatric ophthalmologist at the clinic at the time of study enrollment. Scans should take no longer than 20 seconds each, and ophthalmic exam should take approximately 30 minutes.
  Interventions: Device: Retinal Birefringence Imager

INTERVENTIONS:
Device: Retinal Birefringence Imager — Device is a hand-help object approximately the size of a brick, and is held, by the user, 30cm away from the patient/subject. The subject peers in to an aperture that includes a fixation target that is in the shape of a smiley face. During this time, a ring of LED lights illuminates the eye and captures an image of the retina in approximately 3 seconds. The results instantaneously identify the presence of amblyopia / strabismus.
  Other Names: RBI

SUMMARY:
The purpose of this project is to compare the accuracy of two products at detecting amblyopia and strabismus in children. The devices will be Rebiscan's "blinq" (Pediatric Vision Scanner; PVS) and Rebiscan's RBI (Retinal Birefringence Imager).

DETAILED DESCRIPTION:
Rebiscan is proposing a two-cohort study. The first cohort will include a population enriched for pathology in amblyopia to best assess device sensitivity, while a second cohort will be based in a primary care setting to best assess device specificity. The study will be conducted in busy, ethnically and economically diverse cites affiliated with the Retina Foundation of the Southwest (RFSW) in greater Dallas, TX area. Each child will be screened with Rebiscan's RBI device and it's PVS device in sequence, with results compared to the PVS as well as a comprehensive ophthalmic examination performed by a certified pediatric ophthalmologist in a statistically appropriate subset of screened subjects. Testing times will be assessed to compare the efficiency of the PVS and the RBI screening experiences. The percentage of children successfully completing the screening process will also be measured.

The RBI is expected to identify children with amblyopia and strabismus, without referring children who will not benefit from early treatment

ELIGIBILITY:
Inclusion Criteria:

* Children who present to the participating clinics
* Provide assent
* Guardian provides informed consent

Exclusion Criteria:

- Developmental delay or cognitive deficit

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children between the ages of 2-8, with no gender, race, or ethnicity restricted from enrollment.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Presence of amblyopia / strabismus | 1 single day
  Readouts of RBI device will be compared to clinical examination results

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Birch, PhD, Principal Investigator — Retina Foundation of the Southwest
Locations (1):
- Retina Foundation of the Southwest, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided